CLINICAL TRIAL: NCT01588093
Title: Insulin-like Growth Factor (IGF-I) Induced Muscle Glucose Uptake and Interstitial IGF-1 Concentrations.
Brief Title: IGF-I Induced Muscle Glucose Uptake and Interstitial IGF-I Concentrations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Bang (Other)
Responsible Party: Sponsor-Investigator, Peter Bang, Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: MDIGF-1
Record Dates: First submitted 2012-04-07; First posted 2012-04-30 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — mecasermin; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline (Placebo Comparator)
  Interventions: Drug: 0.9% Saline
- Increlex (Active Comparator)
  Interventions: Drug: Increlex

INTERVENTIONS:
Drug: Increlex — Increlex 120 micrograms/kg body weight single subcutaneous injection
  Arms: Increlex
Drug: 0.9% Saline — Placebo (0,1 ml of 0.9% Saline) single subcutaneous injection
  Arms: Saline

SUMMARY:
Hormonal disturbances in the GH-IGF-I axis are considered important for the deterioration of glycemic control in T1DM particularly in adolescents. In addition it may have direct implications on the development of insulin resistance and long-term complications.

The Investigators hypothesis is that low circulating IGF-I and compensatory hyper-secretion of GH, in the presence of peripheral insulin excess, results in increased local IGF-I expression explaining both the deterioration in metabolic control and the increased risk for microvascular complications. Correction of imbalance in circulating and tissue-specific levels of IGF-I could lead to both better early metabolic control and to prevention of early diabetic complications in type 1 diabetic (T1DM) patients.

Aim of the present study is to validate the microdialysis technique as a useable tool to predict local biological effects of IGF-1 and to understand the pharmacokinetics of local IGF-I actions after sc injection of Increlex in type 1 diabetic patients.

DETAILED DESCRIPTION:
Background:

In healthy subjects, the liver extracts approximately 50 % of insulin. Therefore insulin given subcutaneously results in a relative insulin deficiency in the portal circulation of the liver, and a relative insulin excess in peripheral tissues. In comparison, normal physiological delivery of insulin from the pancreas to the portal circulation, results in markedly higher hepatic insulin exposure. The importance of hepatic insulin exposure for GH induced IGF-I synthesis comes from studies demonstrating that circulating IGF-I levels can be normalized by direct portal insulin infusion (1) or nearly normalized with intra-peritoneal insulin delivery (2). Approximately 80 % of circulating IGF-I is liver derived. Whether the GH induction of IGF-I production in other tissues such as fat, muscle and the growth plate is also insulin dependent has not been studied in humans. While locally produced IGF-I is important for linear growth, circulating IGF-I is essential for insulin sensitivity (3). Portal insulin deficiency results in uncoupling of GH induced IGF-I synthesis and subnormal circulating IGF-I levels in T1DM children with conventional therapy (4).

In newly diagnosed T1DM subcutaneous insulin treatment increases circulating IGF-I (5). The beneficial effects of 12 weeks adjuvant IGF-I treatment on metabolic control was demonstrated in conventionally insulin treated T1DM adolescents (6). There is also strong evidence for the role of IGF-I in the pathogenesis of diabetic kidney disease, atherosclerosis and proliferative retinopathy (7, 8, 9).

Interestingly, recent reports suggest an important role of IGF-I in stimulating beta cell regeneration (10). Thus a role for improvement of IGF-I in prolonging endogenous insulin secretion in the early phase of T1DM disease appears promising.

The Investigators have previously developed a microdialysis approach to measure local IGF-I protein levels from the human muscle tissue. The Investigators were in that study able to show that exercise increases local IGF-I levels. (11, 12) However, no further analysis concerning tissue-specific glucose metabolism was performed.

The Investigators hypothesis is that low circulating IGF-I and compensatory hyper-secretion of GH, in the presence of peripheral insulin excess, results in increased local IGF-I expression explaining both the deterioration in metabolic control and the increased risk for microvascular complications.

In conclusion, correction of imbalance in circulating and tissue-specific levels of IGF-I could lead to both better early metabolic control and to prevention of early diabetic complications in type 1 diabetic (T1DM) patients.

Study Design:

This is a placebo controlled crossover study of the effect of sc IGF-1 (Increlex) administration on glucose infusion rate (whole body glucose utilization) and interstitial muscle IGF-1 concentrations under euglycemic clamp conditions in T1DM adolescents and young adults (18-23 y of age). Each subject is studied twice and randomized to receive IGF-1 (120 μg/ kg, Increlex®, Ipsen) or placebo. Glucose control is optimized by CSII (Continuous Subcutaneus Insulin Infusion) for 2 days and subjects are studied after an overnight fast using a constant low rate insulin infusion to block hepatic glucose production. After a single s.c. bolus of IGF-1, the effects of IGF-1 on the peripheral glucose disposal rate will be assessed based on the rate of a variable glucose infusion. Local muscle IGF-1 measured by microdialysis will be related to the peripheral glucose disposal rate (mainly determined by muscle glucose uptake). Patients with T1DM will be studied for several reasons: 1) They are a target group for long term treatment, 2) They are IGF-I deficient and thus more likely to have a significant effect of sc IGF-I injections, 3) muscle levels may or may not be low.

The following assessments will be performed:

* Height & Weight
* Glucose utilization rate (normoinsulinemic, euglycemic clamp)
* Blood parameters: P-glucose, Growth Hormone (GH), IGF-1, Insulin Like Growth Factor Binding Proteins 1-3 (IGFBP1-3) and Glucagon
* Microdialysis IGF-1

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes duration at least two years and assumed C-peptide negativity
2. Chronological age from 18 to 25 years
3. Tanner stage > 4 (Girls: Tanner B4 or more, Boys: Testis > 15 ml)
4. Levemir or Lantus as basal analogue or CSII
5. IGF-1 < -1.0 SDS and HbA1C < 73 mmol/mol with screening or within past three months
6. Written informed consent

Exclusion Criteria:

1. Development of hypoglycemia that can not be controlled with increased glucose infusion-rate

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Difference in MD (microdialysate) IGF-1 over time (expressed as AUC or peak microdialysate IGF-I) between saline and IGF-I injection. | 0-4 hours from injection

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bang, Professor, Principal Investigator — Karolinska University Hospital, Pediatric Endicrinology Unit, Dept of Women´s and Children´s Health
Locations (1):
- Pediatric Endocrinology Unit, Dept of Women's and Children's Health, Karolinska Institute & University Hospital, Stockholm, Sweden